CLINICAL TRIAL: NCT05720962
Title: The Effect of Continuous Accompanying Support in the Active Phase on Labor Pain, Duration and Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, dilan cömert, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2022/401
Record Dates: First submitted 2023-01-23; First posted 2023-02-09 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Continuous Birth Support
Keywords: continuous birth support; birth time; labor pain; satisfaction
MeSH Terms: conditions — Labor Pain; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: randomized controlled study with two groups as control and experimental group
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The experimental group will be provided with routine midwife support and uninterrupted accompanying support.
  Interventions: Procedure: uninterrupted accompanying support
- control group (No Intervention): Only routine midwife support will be provided to the control group.

INTERVENTIONS:
Procedure: uninterrupted accompanying support — When the participants in the experimental group are taken to the delivery unit, when the neck dilation is 4 cm, a person they want will be taken with them to support them.
  Afterwards, the pain status and satisfaction of the participants will be questioned when it is 4 cm, 6 cm, 8 cm and 10 cm.
  Arms: experimental group

SUMMARY:
This study was planned to determine the effect of continuous accompanying support during the active phase on labor pain, duration and satisfaction.

DETAILED DESCRIPTION:
Participants who comes into childbirth needs the support of people around her in order to cope with the stress, anxiety and labor pain she experiences. This support is the continuous birth support given from the time the participants comes to the hospital until the birth of the baby. Having someone who supports the woman during the birth process will provide a positive birth experience for pregnant women. At the same time, the feeling of pain of the supported woman will be reduced and the delivery time will be shortened.

This randomized controlled study was planned to be performed on primiparous pregnant women between January 2023 and January 2024. The data of the study will be collected with "Personal Information Form", "Visual Analog Scale".

The study was divided into two groups as experimental and control groups. 55 participants in the experiment -55 participants will be randomized to the control group. Participants meeting the inclusion criteria will be asked to rate their pain and satisfaction from 0 to 10 with the VAS 4 cm, 6 cm, 8 cm and fully open. While both groups receive routine midwife support, when the experimental group reaches 4 cm, a person they want will be taken with them and continuous support will be given until there is a dilation of 10 cm.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 years old
* Being literate
* Fluent and speaking Turkish
* Primiparous
* Spontaneous vaginal delivery planned
* At the beginning of the active phase (dilatation 4 cm)
* Pregnant women who agreed to participate in the research

Exclusion Criteria:

* Presence of a health problem in the mother during pregnancy
* At risk of fetal anomaly
* Having multiple pregnancy
* Administering analgesic medication during labor

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 110 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | "through study completion, an average of 1 year"
  It is a reliable and easily applicable scale accepted in the world literature. It is used to measure the values that cannot be measured numerically in the evaluation of the pain intensity and satisfaction of the patients. A minimum of 0 and a maximum of 10 points can be obtained from the scale. Additionally, higher scores indicate higher pain intensity, higher satisfaction.
Personal information form | "through study completion, an average of 1 year".
  It is a form that includes questions that determine socio-demographic characteristics and perception of support. The form also includes questions about the process of the birth period.

CONTACTS AND LOCATIONS:
Overall Officials: Dilan Cömert, Principal Investigator — Msc Midwife
Locations (1):
- Istanbul Universty Cerrahpaşa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No